CLINICAL TRIAL: NCT01911000
Title: Effectiveness and Safety of the Simultaneous Radiotherapy and Hyperthermia After Transarterial Chemoembolization in Hepatocellular Carcinoma Patients Combined With Portal Vein Tumor Thrombosis: Prospective Phase II Trial
Brief Title: Effectiveness and Safety of the Simultaneous Radiotherapy and Hyperthermia After Transarterial Chemoembolization in Hepatocellular Carcinoma Patients Combined With Portal Vein Tumor Thrombosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-06-013-003
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-05

CONDITIONS: Carcinoma. Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

ARMS (1):
- RTHT (Experimental): RT and hyperthermia after TACE in the unresectable HCC patients who combined with PVTT
  Interventions: Radiation: RT and hyperthermia after TACE

INTERVENTIONS:
Radiation: RT and hyperthermia after TACE

SUMMARY:
The presence of portal vein tumor thrombosis (PVTT)in patients with HCC is one of the most significant prognostic factors for poor prognosis, without treatment, their survival is less than 3 months. In the HCC patients who combined with PVTT, RT showed 50% of local control and about 10 months survival duration. Despite the standard treatment of the HCC combined with PVTT is sorafenib, but Korean Liver Cancer Study Group (KLCSG) recommend RT as an option in those patients. Investigators previously reported the retrospective study that the scheduled interval TACE followed by RT for HCC combined with PVTT and 60% of the patients showed objective response without significant elevation of complication. It is reported that hyperthermia considered as the most valuable radiosensitizer in cancer treatment, theoretically. Based on those studies, we start this prospective study to evaluate the objective response and adverse event in the combination treatment of RT and hyperthermia after Transarterial chemoembolization (TACE) in the unresectable HCC patients who combined with PVTT.

DETAILED DESCRIPTION:
1.1 Hepatocellular carcinoma (HCC) and standard treatment HCC is the third most common cause of cancer death globally. It is also the second cause of cancer mortality in Korea, despite the incidence of HCC was fifth. The most important cause of this discrepancy is connected with the fact that the significant portion of the HCC is detected as unresectable status. At the point of HCC diagnosis, only 30% of the patients could receive standard curative treatment, like resection, liver transplantation, and radiofrequency ablation (RFA), TACE has been shown in randomized trials to improve survival compared with symptomatic therapy alone, in the patients without macrovascular involvement, extrahepatic disease and tumor related symptoms. However, in the recent review of TACE, TACE might be contraindicate or not recommended in the patients who showed vascular tumor invasion, more than 10 cm size, poor portal blood flow and/or repeated poor response.

1.2 HCC with PVTT The presence of PVTT in patients with HCC is one of the most significant prognostic factors for poor prognosis, without treatment, their survival is less than 3 months. Recently, Sorafenib, which is one of the target agents, showed survival advantage on unresectable HCC patients in two randomized study. In those study, sorafenib improved approximately three month overall survival increment, however, the median survival duration was only 10.7 months in experiment group (received sorafenib), and even 6.5 months in Asian-Pacific trial. Additionally, the possibility that sorafenib effect could be reduced in the patients had hepatitis B virus (HBV) was suggested in the subgroup analysis.

1.3 Radiation therapy (RT) for the HCC The use of RT in HCC is increased with the radiation technological advances. In the unresectable patients, RT showed 50 to 60% response rate with the dose response relationship. Especially, in the HCC patients who combined with PVTT, RT showed 50% of local control and about 10 months survival duration. Despite the standard treatment of the HCC combined with PVTT is sorafenib, but Korean Liver Cancer Study Group (KLCSG) recommend RT as an option in those patients.

Investigators previously reported the retrospective study that the scheduled interval TACE followed by RT for HCC combined with PVTT and 60% of the patients showed objective response without significant elevation of complication.

1.4 Hyperthermia It is reported that hyperthermia is effective in S phase, Low partial oxygen pressure (pO2), acidic condition, and low perfusion site which are known as radio-resistant. Because of these characteristics, it considered as the most valuable radiosensitizer in cancer treatment, theoretically. Furthermore ,mild hyperthermia (41 to 41.5 ºC) can promote tumor reoxygenation.

1.5 Purpose of the study Based on those studies, we start this prospective study to evaluate the objective response and adverse event in the combination treatment of RT and hyperthermia after TACE in the unresectable HCC patients who combined with PVTT.

2. Hypothesis and sample size Several prospective trials showed 50% to 60% of objective response rate when conventional RT was administered for HCC with PVTT, thus we determined the objective response rate of conventional RT as 60%. We expect additional 20% increase of the local progression free rate than conventional RT when treated with combined RT and hyperthermia for HCC with PVTT.

To determine sample size, we designed to have 80% power to detect an absolute difference of 20% points in objective response rate between combined RT and hyperthermia and conventional RT, with a two-sided alpha level of 0.05. A total of 87 patients are required for this study considering a drop-out rate of 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of HCC by at least one criterion listed below (korean liver cancer study group (KLCSG) guideline 2009) 1.1 Pathologically (histologically or cytologically) proven diagnosis of HCC 1.2 Liver nodule in high risk group 1.2.1 If alpha fetoprotein (AFP) ≥200 ng/mL , ≥ 1 typical HCC enhancing pattern on dynamic contrast enhanced CT or MRI 1.2.2 If AFP<200 ng/mL, ≥2 typical HCC enhancing pattern on dynamic contrast enhanced CT, MRI, and angiography 1.3 ≥ 2 cm nodule in liver cirrhosis (LC), ≥ 1 typical HCC enhancing pattern on dynamic contrast enhanced CT or MRI
2. Patients must have a diagnosis of PVTT 2.1 Early arterial enhancement and delayed washout on multiphasic CT or MRI
3. Eastern cooperative oncology group performance status 0 1 2
4. Age ≥ 20
5. Unsuitable for resection or transplant or RFA
6. Unsuitable for or refractory to TACE or drug eluting beads (DEB)
7. Agreement of study-specific informed consent
8. Assessment by radiation oncologist and medical oncologist or hepatologist within 28 days prior to study entry?
9. Child-Pugh score A-B within 7 days prior to study entry
10. Normal liver (Liver minus gross tumor volume) ≥ 700 cc
11. Blood work requirements

    * Absolute neutrophil count (ANC) ≥ 1,500 /mm3, Platelet ≥ 70,000/mm3, Hgb ≥ 8 g/dl
    * Liver function test (LFT): Total bilirubin<3.0 mg/dL, International normalized ratio(INR) < 1.7, Albumin ≥ 2.8g/dL, Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT)< 6 X normal
    * Serum creatinine < 1.5 X normal, or creatinine clearance ≥ 60 mL/min
12. Male, consent contraception at least 6 months
13. Childbearing potential woman, consent contraception at least 6 months
14. Life expectancy more than 12 weeks
15. Stable breathing more than 5 minutes

Exclusion Criteria:

1. Complete obstruction of main portal vein
2. Pregnant and/or breastfeeding woman
3. Previous upper abdominal RT history
4. Uncontrolled active co-morbidity
5. Another primary cancer history within 2 years
6. Uncontrolled ascites or hepatic encephalopathy
7. Connective tissue disease which known as radiation hypersensitivity
8. Uncontrolled moderate to severe gastroduodenal ulcer or esophagogastric varices

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Hyperthermia effect and averse event in RT for HCC with PVTT | Radiologic response and adverse event will be evaluated at 3 month after treatment.
  Modified response evaluation criteria in solid tumor(mRECIST) will be used. Objective response was defined as complete and partial response. The common terminology criteria for adverse events (CTCAE version 4.0) will be used to evaluate the adverse events.

SECONDARY OUTCOMES:
Hyperthermia effect on local progression free survival rate | The liver CT or MRI will be examined at 3 month after treatment and used to determine the response and presence of progression.
  The liver CT or MRI will be examined at 1, 3 month after treatment, after that 3 month follow-up with above images and used to determine the presence of local progression. Progression free survival will be measured from the date of RT start to the date of local progression recognition or last follow up visit.
To measure the time to local tumor progression | The liver CT or MRI will be examined at 3 month after treatment.
  The liver CT or MRI will be examined at 1, 3 month after treatment, after that 3 month follow-up with above images and used to determine the presence of local progression. Time to local tumor progression will be measured from the date of RT start to the date of local progression recognition.
To measure the overall survival | First follow up will be at 1 month after treatment.
  he follow up will be at 1, 3 month after treatment, after that every 3 month. Overall survival will be measured from the date of RT start to the date of death or last follow up visit.
Quality of life (QoL) change before and after treatment | QoL will be assessed before, 1, 3, 6 months after RT and compared each other.
To validate of the prognostic index of portal vein tumor thrombosis in HCC (PITH) staging system | The liver CT or MRI will be examined at 3 month after treatment
  Overall survival outcome will be used to validate PITH staging system.
To evaluate RT response prediction probability by diffusion-weighted (DW) MRI | DW MRI will be evaluated at 1 month after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Chul Park, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea